CLINICAL TRIAL: NCT04449913
Title: Study of the Longitudinal Changes in Perception and Cognition Occurring During a Meditation Retreat
Brief Title: Changes in Perception and Cognition During a Meditation Retreat
Acronym: LONGIMED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 69HCL20_0003; 2020-A00669-30 (Other: ID-RCB)
Record Dates: First submitted 2020-06-24; First posted 2020-06-29 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Healthy Volunteers
Keywords: Meditation; Emotional Regulation; Metacognitive Awareness; Attention; Mindfulness; Pain; Predictive Coding
MeSH Terms: conditions — Emotional Regulation; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active group (Experimental): 10 days intensive meditation retreat
  Interventions: Behavioral: 10 days intensive meditation retreat
- Control group (Other): Waiting for a 10 days intensive meditation retreat
  Interventions: Behavioral: Waiting for a 10 days intensive meditation retreat

INTERVENTIONS:
Behavioral: 10 days intensive meditation retreat — The intervention consists in a 10 days contemplative retreat, with 6 to 8 hours of sitting and walking meditation per day, and 1 or 2 hours of meditation teachings. The meditation practice will mainly train in mindfulness practice. Mindfulness meditation intends to train attention to detect and regulate afflictive cognitive and emotional patterns. Mindfulness practice requires skills involved in openness to experience, in monitoring the focus of attention and in detecting distraction, disengaging attention from the source of distraction, and flexibly (re)directing and engaging attention to the intended object. A brief introduction to loving-kindness and compassion meditation will also be present throughout the retreat.
  Arms: Active group
Behavioral: Waiting for a 10 days intensive meditation retreat — At the time of measure, participants in this group are waiting to participate to the same meditation retreat as the active group. They may perform their own daily meditation practices as usual.
  Arms: Control group

SUMMARY:
This study aims at assessing neuro-behavioral changes occuring during an intensive ten days meditation retreat. The investigator will study changes in tactile, auditory and pain perceptions as well as changes in cognitive and affective mental contents and their neural markers, as measured by self-reports, EEG event-related potentials, and functional connectivity of resting state fMRI. He will recruit healthy participants with a prior meditation experience. They will be randomly assigned to two groups, one active group who will undergo measurements just before, during and 3 weeks after the retreat. The other group will serve of control for task habituation, control participants will undergo the same measurements, equally spaced in time, but before the retreat. The main hypothesis is that meditation training strengthens meta-awareness, attention capacities resulting in enhanced bodily- and self-awareness during sensory perception and emotion regulation during pain.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 67
* Regular meditation practice (at least 20 minutes 3 times a week) arising from a formal teaching (buddhist tradition, MBSR, mindfulness) for at least one year.
* Having taken part to at least one intensive retreat (more than six hours of sitting meditation a day, during at least two days) in the past.
* Affiliated to french social security
* Motivated to take part in the study
* Having signed an informed consent
* Normal or corrected vision
* Sufficient mastering of French to be able to understand correctly written and auditory instructions

Exclusion Criteria:

* neurological or psychiatric antecedents
* chronical pain or any other medical condition giving rise to acute pain or sensitivity to pain.
* Motor or sensory deficit in the hands
* severe auditory loss
* regularly taking medical drugs acting on the central nervous system
* regularly taking opioids or antidepressant drugs
* alcohol consumption above the safety threshold recognized by the French healthy agency (10 drinks a week, 2 drinks a day, 5 drinks for special occasions)
* drugs consumption (except tabacco) qualified as addictive according to medical criteria (https://www.drogues.gouv.fr/comprendre/l-essentiel-sur-les-addictions/qu-est-ce-qu-une-addiction)
* alcohol or drug consumption the day before or the day of experiment and during the full duration of the retreat
* being pregnant, breastfeading or having given birth less than 6 months ago
* Will be excluded from the fMRI task only, participants presenting contraindication to a MRI scan : being claustrophobic, body mass index over 30, people, having a pacemaker or an insuline pump, metallic prothesis, intracranial clip, neurosensory stimulator, in-body defibrillator, cochlear implants, ocular or brain feromagnetic bodies close to nervous structures, neurosurgery stunts, dental brace.

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2020-10-02 (Actual); Primary Completion 2021-04-10 (Actual); Study Completion 2021-04-10 (Actual)

PRIMARY OUTCOMES:
changes in matched forces (Newtons) during a force-matching task. | 1 or 2 days before the start of the retreat
  Bodily awareness following meditation training could impact the attenuation of real tactile sensations during self-generated touch. Measurement of pressure force will be done through a force-matching paradigm.
changes in matched forces (Newtons) during a force-matching task. | 7 days later
  Bodily awareness following meditation training could impact the attenuation of real tactile sensations during self-generated touch. Measurement of pressure force will be done through a force-matching paradigm.
changes in matched forces (Newtons) during a force-matching task. | at least 3 weeks after the end of the retreat
  Bodily awareness following meditation training could impact the attenuation of real tactile sensations during self-generated touch. Measurement of pressure force will be done through a force-matching paradigm.
changes in EEG an auditory evoked response called the mismatch negativity (microVolt) | 1 or 2 days before the start of the retreat
  Moment-to-moment monitoring following meditation training could downregulate the automatic formation of perceptual habits. Measurement of auditory evoked potentials will be done through Biosemi 64 electrodes EEG net during an auditory oddball task.
changes in EEG an auditory evoked response called the mismatch negativity (microVolt) | 7 days later
  Moment-to-moment monitoring following meditation training could downregulate the automatic formation of perceptual habits. Measurement of auditory evoked potentials will be done through Biosemi 64 electrodes EEG net during an auditory oddball task.
changes in EEG an auditory evoked response called the mismatch negativity (microVolt) | at least 3 weeks after the end of the retreat
  Moment-to-moment monitoring following meditation training could downregulate the automatic formation of perceptual habits. Measurement of auditory evoked potentials will be done through Biosemi 64 electrodes EEG net during an auditory oddball task.
changes in EEG pain-related evoked responses (microVolt) | 1 or 2 days before the start of the retreat
  Moment-to-moment monitoring and emotion regulation following meditation training could downregulate pain catastrophizing. Measurement pain-related evoked potentials will be done through Biosemi 64 electrodes EEG net during a pain characterization task.
changes in EEG pain-related evoked responses (microVolt) | 7 days later
  Moment-to-moment monitoring and emotion regulation following meditation training could downregulate pain catastrophizing. Measurement pain-related evoked potentials will be done through Biosemi 64 electrodes EEG net during a pain characterization task.
changes in EEG pain-related evoked responses (microVolt) | at least 3 weeks after the end of the retreat
  Moment-to-moment monitoring and emotion regulation following meditation training could downregulate pain catastrophizing. Measurement pain-related evoked potentials will be done through Biosemi 64 electrodes EEG net during a pain characterization task.

SECONDARY OUTCOMES:
Changes in perceived pain intensity during a pain paradigm | 1 or 2 days before the start of the retreat
  Moment-to-moment monitoring and emotion regulation following meditation training could regulate the cognitive-affective pain amplificatory processes. Scales ranging from no intensity or unpleasantness, to highest pain intensity or unpleasantness experienced in life will be used during a pain characterization task.
Changes in perceived pain intensity during a pain paradigm | 7 days later
  Moment-to-moment monitoring and emotion regulation following meditation training could regulate the cognitive-affective pain amplificatory processes. Scales ranging from no intensity or unpleasantness, to highest pain intensity or unpleasantness experienced in life will be used during a pain characterization task.
Changes in perceived pain intensity during a pain paradigm | at least 3 weeks after the end of the retreat
  Moment-to-moment monitoring and emotion regulation following meditation training could regulate the cognitive-affective pain amplificatory processes. Scales ranging from no intensity or unpleasantness, to highest pain intensity or unpleasantness experienced in life will be used during a pain characterization task.
Changes in perceived pain unpleasantness during a pain paradigm. | at least 3 weeks after the end of the retreat
  Moment-to-moment monitoring and emotion regulation following meditation training could regulate the cognitive-affective pain amplificatory processes. Scales ranging from no intensity or unpleasantness, to highest pain intensity or unpleasantness experienced in life will be used during a pain characterization task.
Changes in perceived pain unpleasantness during a pain paradigm. | 1 or 2 days before the start of the retreat
  Moment-to-moment monitoring and emotion regulation following meditation training could regulate the cognitive-affective pain amplificatory processes. Scales ranging from no intensity or unpleasantness, to highest pain intensity or unpleasantness experienced in life will be used during a pain characterization task.
Changes in perceived pain unpleasantness during a pain paradigm. | 7 days later
  Moment-to-moment monitoring and emotion regulation following meditation training could regulate the cognitive-affective pain amplificatory processes. Scales ranging from no intensity or unpleasantness, to highest pain intensity or unpleasantness experienced in life will be used during a pain characterization task.
Changes in BOLD functional connectivities at rest and during mindfulness meditation within and between the salience, default mode and executive brain networks | 1 to 7 days before the start of the retreat
  Moment-to-moment monitoring following meditation training could regulate different attention related brain networks. Brain structural anatomy will be recorded in a 3-Tesla fMRI scaner during rest, and BOLD signal activation during rest and meditation states.
Changes in BOLD functional connectivities at rest and during mindfulness meditation within and between the salience, default mode and executive brain networks | 1 to 7 days after the end of the retreat
  Moment-to-moment monitoring following meditation training could regulate different attention related brain networks. Brain structural anatomy will be recorded in a 3-Tesla fMRI scaner during rest, and BOLD signal activation during rest and meditation states.
Changes in BOLD functional connectivities at rest and during mindfulness meditation within and between the salience, default mode and executive brain networks | at least 3 weeks after the end of the retreat
  Moment-to-moment monitoring following meditation training could regulate different attention related brain networks. Brain structural anatomy will be recorded in a 3-Tesla fMRI scaner during rest, and BOLD signal activation during rest and meditation states.
Changes in macroscale functional organization of brain BOLD activity at rest or in meditation | 1 to 7 days before the start of the retreat
  Moment-to-moment monitoring following meditation training could regulate different attention related brain networks. Brain structural anatomy will be recorded in a 3-Tesla fMRI scaner during rest, and BOLD signal activation during rest and meditation states.
Changes in macroscale functional organization of brain BOLD activity in meditation | 1 to 7 days before the start of the retreat
  Moment-to-moment monitoring following meditation training could regulate different attention related brain networks. Brain structural anatomy will be recorded in a 3-Tesla fMRI scaner during rest, and BOLD signal activation during rest and meditation states.
Changes in macroscale functional organization of brain BOLD activity at rest or in meditation | 1 to 7 days after the end of the retreat
  Moment-to-moment monitoring following meditation training could regulate different attention related brain networks. Brain structural anatomy will be recorded in a 3-Tesla fMRI scaner during rest, and BOLD signal activation during rest and meditation states.
Changes in macroscale functional organization of brain BOLD activity in meditation | 1 to 7 days after the end of the retreat
  Moment-to-moment monitoring following meditation training could regulate different attention related brain networks. Brain structural anatomy will be recorded in a 3-Tesla fMRI scaner during rest, and BOLD signal activation during rest and meditation states.
Changes in macroscale functional organization of brain BOLD activity at rest or in meditation | at least 3 weeks after the end of the retreat
  Moment-to-moment monitoring following meditation training could regulate different attention related brain networks. Brain structural anatomy will be recorded in a 3-Tesla fMRI scaner during rest, and BOLD signal activation during rest and meditation states.
Changes in macroscale functional organization of brain BOLD activity in meditation | at least 3 weeks after the end of the retreat
  Moment-to-moment monitoring following meditation training could regulate different attention related brain networks. Brain structural anatomy will be recorded in a 3-Tesla fMRI scaner during rest, and BOLD signal activation during rest and meditation states.
Changes in experiential thought sampling thoughout the meditation retreat. | every day from day 1 to day 10 of the retreat
  Moment-to-moment monitoring of thougts and emotions during intensive meditation training could regulate mind-wandering and mood. Different scales of thoughts content, emotional valence and awareness of them will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Antoine LUTZ, PhD, Principal Investigator — Centre de recherche de Neurosciences de Lyon (CRNL)
Locations (1):
- Centre de Recherche en Neuroscience de Lyon, Bron, France